CLINICAL TRIAL: NCT04945330
Title: Special Drug Use Investigation for Larotrectinib
Brief Title: NTRK Gene Fusion - Positive Advanced or Recurrent Solid Tumors, a Rare Cancer Caused by Specific Changes in the Genes
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21793
Record Dates: First submitted 2021-06-20; First posted 2021-06-30 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Advanced or Recurrent Solid Tumor Harboring an NTRK Gene Fusion
MeSH Terms: interventions — larotrectinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Gastrointestinal (GI): Participants with GI cancer.
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Head and neck (H&N): Participants with H&N cancer.
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Lung: Participants with lung cancer.
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Soft tissue sarcoma (STS): Participants with STS cancer.
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Primary central nervous system (CNS): Participants with CNS cancer.
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Melanoma: Participants with Melanoma cancer.
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Pediatrics
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)
- Others
  Interventions: Drug: Larotrectinib (Vitrakvi, BAY2757556)

INTERVENTIONS:
Drug: Larotrectinib (Vitrakvi, BAY2757556) — Follow clinical practice

SUMMARY:
Researchers want to learn more about the use of larotrectinib as a real-world treatment for tropomyosin receptor kinase fusion cancer, also called TRK fusion cancer.

In people with TRK fusion cancer, a gene called neurotrophic TRK, (NTRK) joins or "fuses" with another gene. This creates a protein known as a fusion protein, which can cause cancer cells to grow. The study treatment, larotrectinib, is already available for doctors to prescribe to patients with TRK fusion cancer. Larotrectinib works by blocking TRK genes in cancer cells which helps stop the cancer from growing.

In this study, the researchers want to learn more about the safety and effectiveness of larotrectinib in adults and children with advanced or recurrent TRK fusion cancer. This means that their cancer has spread from where it started to other areas of the body, or the cancer has come back after a period of time. To answer this question, the researchers will collect information from patients who are taking larotrectinib as prescribed by their doctors. The researchers will learn what adverse events the patients are having. An adverse event is any medical problem that a patient has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

The study will include patients of all ages with TRK fusion cancer.

In this study, there will be no required tests or visits to a study site. Instead, the researchers will collect information from:

* the patients' medical records
* interviews with the patients or their parents or guardians
* the patients' visits to their doctor as part of their usual care The researchers will collect information about the adults for up to about 2 years and about the children for up to about 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated with larotrectinib or decided to be treated with larotrectinib, under routine clinical practice.

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric (from birth to 18 year old) patients treated with larotrectinib.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of treatment emergent adverse events (TEAEs) | Approximate 8 years
Frequency of TEAEs | Approximate 8 years
Seriousness of TEAEs | Approximate 8 years
Outcome of TEAEs | Approximate 8 years
Causality assessment of TEAEs | Approximate 8 years

SECONDARY OUTCOMES:
Overall response rate (ORR), based on investigator assessment preferably using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or Response Assessment in Neuro-Oncology (RANO) as appropriate by local investigator assessment | Approximate 8 years
Disease control rate (DCR) | Approximate 8 years
Duration of response (DOR) | Approximate 8 years
Time to response (TTR) | Approximate 8 years
Progression-free survival (PFS) | Approximate 8 years
Overall survival (OS) | Approximate 8 years
Total dose | Approximate 8 years
Starting and ending dose | Approximate 8 years
Dose modification during treatment | Approximate 8 years
Duration of treatment (DOT) | Approximate 8 years
Baseline characteristics | Approximate 8 years
  Including but not limited to: age, NTRK gene, NTRK gene partner, prior therapy (type, number of lines of therapy), other.
Neurological examination (normal/abnormal) | Approximate 8 years
Change in height from baseline by visit | Approximate 8 years
Change in weight from baseline by visit | Approximate 8 years
Developmental milestones abnormalities (normal/abnormal) | Approximate 8 years

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.